CLINICAL TRIAL: NCT00557791
Title: A Phase 3, Randomized, Double-masked, Parallel-assignment and Dose-finding Study of Intravitreal Bevasiranib Sodium, Administered Every 8 Weeks as Maintenance Therapy Following Three Injections of Lucentis® Compared With Lucentis® Monotherapy Every 4 Weeks in Patients With Exudative Age-Related Macular Degeneration (AMD).
Brief Title: Safety & Efficacy Study Evaluating the Combination of Bevasiranib & Lucentis Therapy in Wet AMD (CARBON)
Acronym: CARBON
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study never initiated
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Naveed Shams, Opko Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACU302
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2011-02

CONDITIONS: Age Related Macular Degeneration
Keywords: AMD; ARMD; Exudative Macular Degeneration; Bevasiranib; siRNA
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration | interventions — bevasiranib; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Active Comparator): Lucentis® (0.5 mg) every 4 weeks.
  Interventions: Drug: ranibizumab
- B (Experimental): Bevasiranib (1.0 mg) every 8 weeks beginning at week 12, after pre-treatment with 3 injections of Lucentis® and initial priming doses of bevasiranib at weeks 2 & 6.
  Interventions: Drug: Bevasiranib
- C (Experimental): Bevasiranib (2.0 mg) every 8 weeks beginning at week 12, after pre-treatment with 3 injections of Lucentis® and initial priming doses of bevasiranib at weeks 2 & 6.
  Interventions: Drug: Bevasiranib
- D (Experimental): Bevasiranib (2.5 mg) every 8 weeks beginning at week 12, after pre-treatment with 3 injections of Lucentis® and initial priming doses of bevasiranib at weeks 2 & 6.
  Interventions: Drug: Bevasiranib

INTERVENTIONS:
Drug: Bevasiranib — Three doses (1.0mg, 2.0mg, 2.5mg) of bevasiranib administered intravitreally every 8 weeks
  Arms: B; C; D
Drug: ranibizumab — Lucentis® (0.5 mg) administered intravitreally every 4 weeks.
  Other Names: Lucentis®
  Arms: A

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of three doses of intravitreal bevasiranib sodium as maintenance therapy for Age-Related Macular Degeneration following initiation of anti-VEGF therapy with three doses of Lucentis®.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be age 50 years or older
* Patients must have predominantly classic, minimally classic or occult with no classic lesions secondary to Age Related Macular Degeneration.
* The study eye must have ETDRS best corrected visual acuity of 69 to 24 letters (20/40 to 20/320 Snellen equivalent).
* Patients must be willing and able to return for scheduled monthly follow-up visits for two-years.

Exclusion Criteria:

* Prior pharmacologic treatment for AMD in the study (patients can not have previously received Avastin®/Lucentis®, Macugen®, or any other anti-VEGF agents, steroid treatments, PDT, radiation treatment, or any experimental therapies for AMD in the study eye)
* Any intraocular surgery of the study eye within 12 weeks of screening
* Previous posterior vitrectomy of the study eye
* Advanced glaucoma or intraocular pressure above 22 mm Hg in the study eye despite treatment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy measure: The proportion of patients at week 60 in each group with a successful visual acuity outcome (as defined as avoidance of a 3, or more, line loss in vision). | 60 weeks

SECONDARY OUTCOMES:
Time from tx initiation to 1st use of rescue | 60 weeks
Distribution of change in VA from baseline to 60 weeks | 60 weeks
Proportion of patients at week 60 with a 3, or more, line gain in vision | 60 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Shams, MD, Study Director — SVP at Opko Health